CLINICAL TRIAL: NCT05129787
Title: A Randomized Controlled Trial of Needle Ablation With 3D Verification vs Surgical Resection of Colorectal Cancer Liver Metastases
Brief Title: Ablation vs Resection of Colorectal Cancer Liver Metastases
Acronym: NEW-COMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Åsmund Avdem Fretland, Consultant HPB surgeon, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REK255384
Record Dates: First submitted 2021-11-02; First posted 2021-11-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Masking will be performed by large drapings on wounds and masking of operation notes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical resection (Active Comparator): Liver resection
  Interventions: Procedure: Surgical resection
- Thermal ablation (Experimental): Thermal ablation (Microwave or radiofrequency)
  Interventions: Procedure: Thermal ablation

INTERVENTIONS:
Procedure: Surgical resection — Resection of metastasis
  Arms: Surgical resection
Procedure: Thermal ablation — Ablation of metastasis
  Arms: Thermal ablation

SUMMARY:
230 patients with colorectal cancer liver metastases will be randomly assigned to resection or thermal ablation.

DETAILED DESCRIPTION:
Rationale: The use of thermal ablation of liver tumors is rapidly increasing. This is despite a lack of high-level evidence of the oncologic efficacy of ablation. Ablation is most often used in cases where resection is not possible, but as the technique has improved it is increasingly used as a substitute for resection. A majority of studies on ablation are hampered by selection bias. Selection bias can only be overcome in a randomized controlled trial.

Primary objective:

To compare rates of local tumor progression within 12 months in patients randomly assigned to thermal ablation or surgical resection of colorectal liver metastases.

Secondary objectives:

* To establish a pipeline for immediate three-dimensional verification of the ablated zone following thermal ablation of liver metastases.
* To compare health related quality of life in patients randomly assigned to thermal ablation or surgical resection of colorectal liver metastases.
* To perform a cost-effectiveness analysis (Cost per quality adjusted life year) of thermal ablation and resection of colorectal liver metastases.
* To compare disease-free and overall survival in in patients randomly assigned to thermal ablation or surgical resection of colorectal liver metastases.
* To evaluate the hemodynamic response to thermal ablation and laparoscopic resection of liver tumors.

Study design:

A randomized, controlled, multicenter, double-blinded non-inferiority trial.

Study population:

Two groups of 115 patients (230 in total) with colorectal liver metastasis eligible for radical treatment using EITHER resection OR ablation (not a combination).

Intervention:

Ablation of colorectal liver metastases

Control:

Resection of colorectal liver metastases

Main study parameters/endpoints:

The primary endpoint of the study is local recurrence of cancer at 12 months. Secondary endpoints include overall survival, disease free survival, health related quality of life, postoperative pain, complications, hospital stay and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified colorectal cancer
* Colorectal liver metastases (proven or suspected) eligible for radical treatment using EITHER resection OR ablation (not a combination), as decided by the liver MDT meeting at the study center
* The patient is fit to undergo both resection and ablation of all liver metastases
* Size of largest lesion up to and including 30 mm
* In case of solitary metastasis, resection plan includes resection of ≤ 2 anatomical segments.
* In case of multiple metastases in one continuous resection, resection plan can include ≤ 4 anatomical segments (including hemihepatectomy)
* ≤ 5 tumors to be treated in one procedure
* Primary tumor either resected (primary first) or with a plan for curative treatment (liver first).

Exclusion Criteria:

• More than 3 lung metastases where 1 is >10mm, or 1 lung metastasis >15 mm (OR: unresectable lung metastases as decided by the lung MDT meeting)

* Presence of extrahepatic, extrapulmonary metastases.
* Surgical indication for removal of enlarged lymph nodes in the hepatic hilum. (Enlarged lymph nodes without indication of removal are not considered an exclusion criterium)
* Tumor closer than 10 mm to right/left main bile duct
* Suspected tumor infiltration to adjacent organs
* Progression (as of RECIST [18]) on 2nd line chemotherapy
* Previous inclusion in this trial
* Not eligible for workup according to study criteria
* Contraindication to contrast enhanced CT scan
* Manifest liver cirrhosis
* Pregnancy
* ECOG performance status ≥3
* Simultaneous resection of primary tumor or any other concomitant surgical procedure
* Any other reason why, in the investigator's opinion, the patient should not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2030-10-23 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression | 12 months
  Local tumor progression at site of treatment

SECONDARY OUTCOMES:
Overall survival | 60 months
  Overall survival following treatment
Overall survival (secondary analysis) | 60 months
  A secondary analysis will be performed on a oncologically more homogenous group of patients that fulfil the following requirements: a) no previous surgical procedure on the liver, b) no extrahepatic metastases, and c) that had their primary tumor resected
Disease free survival | 60 months
  DFS
Postoperative complications | 30 days
  Morbidity
Health related quality of life | 12 months
  HRQoL is measured using SF-36
Cost-Effectiveness | 12 months
  An analysis of cost will be performed to assess cost-effectiveness
Hemodynamic response | 7 days
  The hemodynamic response to the two interventions will be recorded and compared
Ventilation methods | 1 day
  The intraoperative movement of the liver will be measured using different ventilation methods (one lung ventilation, jet ventilation, gentle double lung ventilation). The movement of the liver during the different ventilation methods will be assessed in cm.
Cerebral flow | 1 day
  Intraoperative cerebral blood flow will be measured and related to cardiac output and other hemodynamic measures. Micro bubbles caused by the treatment will be visualized using ultrasonography.
Inflammatory response | 7 days
  The inflammatory response (cytokines, complement, catecholamines) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Edwin, Professor, Study Director — Head of clinical research, The Intervention Centre, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Department of Gastrointestinal surgery, The National Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD maybe shared pending approval from local data protection officer
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3-5 years
Access Criteria: Upon contact to PI

REFERENCES:
- [Derived] Hansen IS, Lappen KR, Brudvik KW, Rosok BI, Bjork I, Ostergaard D, Andersen MH, Pelanis E, Espinoza AW, Halvorsen PS, Yaqub S, Lassen K, von Gohren Edwin B, Syversveen T, Fretland AA. A Randomized Controlled Trial of Resection Versus Thermal Ablation of Colorectal Cancer Liver Metastases (New Comet): Study Protocol. Ann Surg Oncol. 2025 Aug 26;32(12):9146-53. doi: 10.1245/s10434-025-17984-5. Online ahead of print. PMID 40858956